CLINICAL TRIAL: NCT02925468
Title: Orthodontic Reduction of an Increased Overbite in Adolescents - the Mechanism and Rate of Occlusal Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Evelyn Dunbar, Principal Investigator, NHS Tayside
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016DE02
Record Dates: First submitted 2016-09-22; First posted 2016-10-05 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Increased Overbite
Keywords: orthodontics
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): A standard initial lateral cephalogram radiograph will be taken of all subjects, unless this is already available within the specified age range. An intra-oral scanner will be used to accurately record the occlusal relationships prior to insertion of the fixed anterior bite plane (bite turbos) (T0) and repeated immediately after placement (T1). Each subject will then be re-scanned on a six weekly basis for a period of six months (T2-T5). Conventional clinical photographs and three-dimensional stereophotogrammetry will be used to assess the vertical facial relationships at T0-T5. A further lateral cephalogram radiograph will be taken at T5.
  Interventions: Device: Bite turbo
- Control group (No Intervention): A control group of subjects from the treatment waiting list who meet the inclusion criteria will be used. An intra-oral scanner will record the baseline occlusal relationship (T0) and will be repeated after six months (T5). The control group will also have a standard pre-treatment lateral cephalogram radiograph taken, as well as conventional and three-dimensional stereophotogrammetry at baseline (T0) and after six months (T5). This will allow changes resulting from growth to be assessed whilst no active orthodontic treatment has taken place.

INTERVENTIONS:
Device: Bite turbo — In this study the nature and speed of adaptation of the occlusal changes following insertion of an anterior bite plane (bite turbos) for the reduction of a deep overbite in growing patients will be investigated.
  Other Names: Ormco Europe 350-0000
  Arms: Intervention group

SUMMARY:
The correction of a deep overbite is assumed to involve incisor intrusion and the extrusion or eruption of premolars and molars. The latter is also assumed to be the major contributor for growing patients where the vertical facial growth increase accommodates for the additional eruption of posterior teeth with anterior bite plane appliances.

In this study the nature and rate of adaptation of the occlusal changes following insertion of a fixed anterior bite plane for the reduction of a deep overbite in growing patients will be investigated.

DETAILED DESCRIPTION:
All subjects who meet the inclusion criteria will be informed of the study and written consent sought for their participation. Subjects will be recruited from the new patient clinics and routine treatment waiting list. A standard initial lateral cephalogram will be taken of all subjects, unless this is already available within the specified age range. Active growth will be determined using the Bacetti CVM method. For the Intervention group - an intra-oral scanner will be used to accurately record the occlusal relationships prior to insertion of the fixed anterior bite plane (T0) and repeated immediately after placement (T1). Each subject will then be re-scanned on a six weekly basis for a period of six months (T2-T5). Conventional clinical photographs and three-dimensional stereophotogrammetry will be used to assess the vertical facial relationships at T0-T5. A further lateral cephalogram will be taken at T5 to assess for skeletal change and assess for evidence of intrusion and eruption as well as determine if there has been an alteration in incisor inclination.

A control group of subjects from the treatment waiting list who meet the inclusion criteria will be used. An intra-oral scanner will record the baseline occlusal relationship (T0) and will be repeated after six months (T5). The control group will also have a standard pre-treatment lateral cephalogram taken, as well as conventional and three-dimensional stereophotogrammetry at baseline (T0) and after six months (T5). This will allow changes resulting from growth to be assessed whilst no active orthodontic treatment has taken place.

The primary outcomes to be assessed will be the nature of the change in occlusal-vertical dimension and the rate of occlusal adaptation in relation to facial growth changes. The intra-oral scans and photographs will be analysed using three-dimensional technology to determine the immediate change and any resultant occlusal adaptation and change in lower face height on a six weekly basis for six months.

All subjects and guardians in the intervention group will be asked to complete a short questionnaire immediately after visits T1 and T5. This will assess their experience of the 3-D scanning and bite planes (if applicable). We will also assess their knowledge of overbite definition, process of overbite reduction and effects of an increased overbite on oral health. The control group will be asked to complete the same questionnaire at T0.

The economic impact of managing the increased overbite as an initial phase of treatment versus single phase comprehensive treatment will be investigated. A cost analysis will be performed to investigate any economic difference in using bite turbos versus a removable appliance to reduce the overbite.

ELIGIBILITY:
Inclusion Criteria:

* Class II division 2 malocclusion
* No history of active orthodontic treatment
* Increased overbite (greater than one third lower incisal coverage)
* Age 9-16

Exclusion Criteria:

* Restorations on the palatal surface of the maxillary incisors
* Increased overjet where the lower incisor edge occludes distal to the cingulum of the upper incisor
* Profound hypodontia (>1 missing tooth per quadrant)
* Subjects beyond pubertal growth stage
* Suspected or identifiable syndromes
* Subjects with cleft lip and palate
* Growth anomalies or taking growth accelerating/ inhibiting medication

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
The rate of occlusal reestablishment (measured as first molar contact) following insertion of fixed anterior bite planes (measured in weeks) | Measured 6-weekly for a period of 6 months (T0-T5)
  An intra-oral scanner will allow detailed analysis of the occlusal changes following insertion of fixed anterior bite planes. Participants will be re-scanned every 6 weeks for a period of 6 months to determine if and when first molar contact is re-established.

SECONDARY OUTCOMES:
The acceptability of fixed anterior bite planes and intra-oral scanning in adolescents (questionnaire) | 6 months
  A questionnaire will be used in the intervention group after 6 months to determine the acceptability of the fixed bite planes
If treatment with bite planes increases participants knowledge of overbite reduction and relation to oral health/ orthodontic treatment (questionnaire) | 6 months
  Questionnaires will be used at T0 and T5 (in the intervention group) to assess participants knowledge of overbite reduction and its impact on dental health.
Economic impact of using fixed bite planes as an alternative to a removable appliance (measured in pounds sterling) | 6 months
  An estimate will be made of the cost of providing the fixed bite planes compared to the standard method of overbite reduction using a removable appliance
The nature of occlusal changes following insertion of fixed anterior bite planes | Measured 6-weekly for a period of 6 months (T0-T5)
  An intra-oral scanner will allow detailed analysis of what occlusal changes occur (eruption/intrusion) following insertion of fixed anterior bite planes

CONTACTS AND LOCATIONS:
Overall Officials: Grant McIntyre, Principal Investigator — NHS Tayside
Locations (1):
- Dundee Dental Hospital, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided